CLINICAL TRIAL: NCT07260396
Title: Comparison of the Cutaneous Sensory Block Coverage of Surgical Incisions and Clinical Effectiveness of TAP and Rectus Sheath Blocks in Total Abdominal Hysterectomies Performed With a Pfannenstiel Incision: A Prospective Observational Study
Brief Title: Comparison of Sensory Block Coverage and Clinical Effectiveness of TAP and Rectus Sheath Blocks in Pfannenstiel Incisions
Status: Not yet recruiting | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: GOKAEK 2025/20/18
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Pain Management; Hysterectomy
Keywords: Regional Anesthesia; Postoperative Pain; Cutaneous Sensory Mapping
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Transversus Abdominis Plane Block (TAPB): Patients who received an ultrasound-guided bilateral Transversus Abdominis Plane Block during the preoperative period.
  Interventions: Procedure: Group Transversus Abdominis Plane Block
- Group Rectus Sheath Block (RSB): Patients who received an ultrasound-guided bilateral Rectus Sheath Block during the preoperative period.
  Interventions: Procedure: Group Rectus Sheath Block

INTERVENTIONS:
Procedure: Group Transversus Abdominis Plane Block — Patients will receive a bilateral transversus abdominis plane block preoperatively under ultrasound guidance.
  Bilateral blocks will be performed using 0.25% bupivacaine (25 mL per side, total 50 mL). Sensory block areas will be evaluated using pinprick at predefined time points. Additionally, patients will be provided with a PCA device, and morphine consumption as well as NRS pain scores will be monitored at regular intervals.
  Groups: Group Transversus Abdominis Plane Block (TAPB)
Procedure: Group Rectus Sheath Block — Patients will receive a bilateral rectus sheath block preoperatively under ultrasound guidance.
  Bilateral blocks will be performed using 0.25% bupivacaine (25 mL per side, total 50 mL). Sensory block areas will be evaluated using pinprick at predefined time points. Additionally, patients will be provided with a PCA device, and morphine consumption as well as NRS pain scores will be monitored at regular intervals.
  Groups: Group Rectus Sheath Block (RSB)

SUMMARY:
Hysterectomy is one of the most common major gynecologic surgeries performed for various indications, and hundreds of thousands of procedures are carried out annually, particularly in developed countries. In total abdominal hysterectomies, the Pfannenstiel incision is frequently preferred due to its advantages in terms of aesthetics, functionality, and postoperative recovery. However, this incision can cause significant postoperative pain because of the extensive cutaneous innervation of the lower abdominal wall. This pain may delay early mobilization and negatively affect patient comfort and satisfaction.

As part of multimodal analgesia strategies, regional anesthesia techniques are widely used in such surgeries to reduce opioid consumption and enhance analgesic efficacy. In this context, the Transversus Abdominis Plane (TAP) block and the Rectus Sheath Block (RSB) are among the effective techniques targeting the anterior abdominal wall, and various studies have investigated their spread patterns and clinical outcomes. However, data on the extent to which these blocks provide cutaneous sensory coverage of the Pfannenstiel incision remain limited, and direct comparative mapping studies are scarce in the literature.

For patients undergoing hysterectomy, regional anesthesia techniques are commonly applied perioperatively either as a single technique or in combination for pain management, with TAP and RSB being the most frequently used modalities. In addition, patient-controlled analgesia (PCA) devices are routinely employed as a component of multimodal pain management in this population.

The aim of this study is to comparatively evaluate the cutaneous sensory block areas produced by the TAP and RSB regional anesthesia techniques, their rates of coverage of the Pfannenstiel incision, and their clinical effectiveness.

DETAILED DESCRIPTION:
Inadequate pain control after hysterectomy is associated with prolonged hospital stay, delayed recovery, decreased quality of life, and reduced patient satisfaction. Therefore, multimodal analgesia strategies that provide high analgesic efficacy with a low side-effect profile are essential in these patients during the postoperative period. Effective postoperative analgesia may also reduce the risk of developing chronic pain after hysterectomy. Although opioids are often routinely used in the postoperative period, their widespread use may lead to adverse effects such as nausea and vomiting, constipation, pruritus, urinary retention, respiratory depression, and, in the long term, an increased risk of misuse.

In our clinic, regional anesthesia techniques under ultrasound guidance are routinely administered by experienced anesthesiologists-either as single techniques or in combination-for perioperative pain management in patients undergoing hysterectomy. In addition, patient-controlled analgesia (PCA) devices are used as part of multimodal pain management.

This study was designed as an observational study. It aims to comparatively evaluate the cutaneous sensory block areas produced by bilateral Transversus Abdominis Plane (TAP) block and bilateral Rectus Sheath Block (RSB) in patients undergoing elective total abdominal hysterectomy with a Pfannenstiel incision under general anesthesia, focusing on the extent to which these regional anesthesia techniques cover the Pfannenstiel incision and their clinical effectiveness.

Among the patients who receive either of these techniques, written informed consent will be obtained, and sensory anesthesia will be evaluated at the 45th minute using the pinprick test. The sensory borders identified during the assessment will be marked on the patient's abdomen, after which an acetate sheet will be placed over the abdomen to transfer the anatomical projection of these borders. Additionally, anterior abdominal reference landmarks specific to each patient (xiphoid process, costal margin, anterior axillary line, iliac crest, inguinal ligament, and symphysis pubis) will be marked on the acetate sheet. Before the surgery begins, the Pfannenstiel incision planned by the surgeon will be drawn on the patient and transferred onto the acetate sheet.

Each acetate template will then be digitized, and the percentage of Pfannenstiel incision coverage by the cutaneous sensory block area produced by the regional anesthesia technique will be calculated using ImageJ software. Furthermore, the percentage of the anterior abdominal wall covered by the bilaterally applied regional anesthesia technique will be calculated separately for each patient.

Postoperatively, patients' pain scores will be recorded at 1, 3, 6, 12, 18, and 24 hours using the Numerical Rating Scale (NRS), both at rest and during coughing. Total analgesic consumption from the PCA device will also be documented at the same time intervals. At the end of the 24th hour, all patients will be assessed using the Quality of Recovery-15 (QoR-15) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II-III
* Patients scheduled for elective total abdominal hysterectomy under general anesthesia and who have received either a preoperative rectus sheath block or a transversus abdominis plane block
* Aged 18-70 years
* Patients who agree to participate in the study and provide written informed consent

Exclusion Criteria:

* Patients who refuse to participate
* Patients who have not received any regional anesthesia technique
* ASA physical status IV
* Patients in whom unilateral or bilateral sensory spread is not observed following the bilaterally applied regional anesthesia technique
* Patients who are uncooperative or have cognitive impairment or dementia
* Patients with psychiatric disorders such as depression, mania, or schizophrenia, or those using antipsychotic medications for more than 4 weeks

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients undergoing total abdominal hysterectomy with a Pfannenstiel incision will be included in the study.
Study Population: Patients scheduled for total abdominal hysterectomy with a Pfannenstiel incision and receiving regional anesthesia as part of their perioperative analgesia management will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Calculation of the coverage rates of the Pfannenstiel incision by the cutaneous sensory block areas generated by the transversus abdominis plane block and the rectus sheath block. | 45 minutes after block application

SECONDARY OUTCOMES:
Calculation of the coverage rates of the anterior abdomen by the cutaneous sensory block areas generated by the transversus abdominis plane block and the rectus sheath block. | 45 minutes after block application
Comparison of 24-hour morphine consumption between the two groups. | First 24 postoperative hours
Comparison of Numerical Rating Scale (NRS) scores between the two groups. | Postoperative 1, 3, 6, 12, 18, and 24. hours
Comparison of Quality of Recovery-15 (QoR-15) scores between the two groups. | 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Akdeniz, Study Director — Samsun University

REFERENCES:
- [Background] Aoyama Y, Sakura S, Abe S, Wada M, Saito Y. Analgesic effects and distribution of cutaneous sensory blockade of quadratus lumborum block type 2 and posterior transversus abdominis plane block: an observational comparative study. Korean J Anesthesiol. 2020 Aug;73(4):326-333. doi: 10.4097/kja.19404. Epub 2020 Jan 31. PMID 32008278
- [Background] Abuelghar WM, El-Bishry G, Emam LH. Caesarean deliveries by Pfannenstiel versus Joel-Cohen incision: A randomised controlled trial. J Turk Ger Gynecol Assoc. 2013 Dec 1;14(4):194-200. doi: 10.5152/jtgga.2013.75725. eCollection 2013. PMID 24592105
- [Background] Pickett CM, Seeratan DD, Mol BWJ, Nieboer TE, Johnson N, Bonestroo T, Aarts JW. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2023 Aug 29;8(8):CD003677. doi: 10.1002/14651858.CD003677.pub6. PMID 37642285